CLINICAL TRIAL: NCT02952781
Title: Comparison of Continuous Sternal ECG Patch Monitors (Carnation and Zio) Trial
Status: Completed | Type: Observational
Sponsor: EvergreenHealth (Other)
Responsible Party: Sponsor
Other Study IDs: CZ2016
Record Dates: First submitted 2016-10-13; First posted 2016-11-02 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Syncope; Presyncope; Atrial Fibrillation; Supraventricular Tachycardia
Keywords: ECG Monitoring; Palpitations
MeSH Terms: conditions — Syncope; Atrial Fibrillation; Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EKG Patch monitors (Zio and Carnation) — Each patient will be provided with both a Zio-XT Patch monitoring system and the CAM system and will be instructed to wear both simultaneously for 7 days.

SUMMARY:
The purpose of this research is to test the clinical value of a new P-wave sensitive recording vector compared to a standard ECG limb lead II vector from similar easy-to-use long-term cardiac rhythm monitoring patch systems, the Carnation TM Ambulatory Monitoring (CAM) System and the Zio-XT iRhythm. The P-wave is a critical aspect of the electrocardiogram. The purpose of this study is to see if the P-wave centric focus of the CAM system improves arrhythmia diagnosis.

DETAILED DESCRIPTION:
This study is intended to compare the new Carnation patch monitoring system with the Zio patch, which represents the current standard for continuous recording of the ECG over extended periods. The primary endpoint for this comparison will be diagnostic yield with secondary endpoints being ease of use and comfort.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Written informed consent
* Patients with one or more of the following:

  * Syncope of uncertain etiology; or
  * Pre-syncope of uncertain etiology; or
  * Palpitations of uncertain etiology; or
  * Management of known AF/SVT patients

Exclusion Criteria:

* Any dermatitis or infected skin over the sternum (Carnation patch) or left upper anterior thorax (Zio patch).
* A sternal or thoracic incision that extends under the patch within 3 months from the date of enrollment.
* Cognitive deficits that would interfere with the subject's ability to give informed consent or perform study testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac patients followed at the study site's location.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
ECG signal quality | 7 days
  ECG signal quality = scoring the ability of each system to record electrical activity from the atrium (P-waves). The Physician Event Committee will independently score the P-waves from all recordings.

SECONDARY OUTCOMES:
Skin comfort or discomfort: Was skin irritated? | 7 days
  User will rate skin comfort on pre-determined scale: None, Mild, Moderate, Severe.
Device Comfort | 7 days
  Was device comfortable to wear? User will rate on a predetermined scale: Very Uncomfortable, Mildly Uncomfortable, Comfortable.
Device Stability and Contact | 7 days
  Did the device stay in place in the chest location where it was attached for the time period indicated? Clinician will evaluate visually, and rate on a predetermined scale: Yes, No.
Diagnostic Yield | 7 days
  Diagnostic Yield: proportion of patients for whom an arrhythmogenic source of symptoms is established or eliminated as a diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Vossler, MD, Principal Investigator — Evergreenhealth Heart and Vascular Care
Locations (1):
- EvergreenHealth Heart and Vascular Care, Kirkland, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bass EB, Curtiss EI, Arena VC, Hanusa BH, Cecchetti A, Karpf M, Kapoor WN. The duration of Holter monitoring in patients with syncope. Is 24 hours enough? Arch Intern Med. 1990 May;150(5):1073-8. PMID 2331188
- [Result] Clinical value of vectorcardiography, Holter monitoring and quantitative electrocardiology. Belgian Society of Cardiology. Working Group on Electrocardiology, Exercise Testing and Cardiac Rehabilitation. Acta Cardiol. 2000 Jun;55(3):157-62. doi: 10.2143/AC.55.3.2005733. PMID 10902039
- [Result] Bell C, Kapral M. Use of ambulatory electrocardiography for the detection of paroxysmal atrial fibrillation in patients with stroke. Canadian Task Force on Preventive Health Care. Can J Neurol Sci. 2000 Feb;27(1):25-31. doi: 10.1017/s0317167100051933. PMID 10676584
- [Result] Brown AP, Dawkins KD, Davies JG. Detection of arrhythmias: use of a patient-activated ambulatory electrocardiogram device with a solid-state memory loop. Br Heart J. 1987 Sep;58(3):251-3. doi: 10.1136/hrt.58.3.251. PMID 3663425
- [Result] Calkins H, Byrne M, el-Atassi R, Kalbfleisch S, Langberg JJ, Morady F. The economic burden of unrecognized vasodepressor syncope. Am J Med. 1993 Nov;95(5):473-9. doi: 10.1016/0002-9343(93)90329-n. PMID 8238063
- [Result] Clark PI, Glasser SP, Spoto E Jr. Arrhythmias detected by ambulatory monitoring. Lack of correlation with symptoms of dizziness and syncope. Chest. 1980 Jun;77(6):722-5. doi: 10.1378/chest.77.6.722. PMID 7398383
- [Result] Cumbee SR, Pryor RE, Linzer M. Cardiac loop ECG recording: a new noninvasive diagnostic test in recurrent syncope. South Med J. 1990 Jan;83(1):39-43. doi: 10.1097/00007611-199001000-00013. PMID 2300833